CLINICAL TRIAL: NCT04811261
Title: u-STOP LVAD Bleed: Utilization of Umbilical Cord Lining Stem Cells (ULSCs) To Prevent Left Ventricular Assist Device (LVAD) Associated Angiodysplastic Bleeding
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: u-STOP LVAD Bleed; IRB202100247 (Other: UF IRB-01); OCR40194 (Other: UF OnCore)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Angiodysplastic Bleeding

STUDY DESIGN:
Intervention Model Description: Subjects will be entered into a 3+3 dose escalation study, a standard design for initial trials to evaluate tolerability of a therapeutic agent and identify a maximal tolerated dose if indeed toxicities are identified in the pre-specified dosing range.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3+3 dose escalation (Experimental): The first 3 subjects' patients will be administered 50 x 10^6 ULSCs reconstituted in PBS with 1% human serum albumin in a volume of 250 ml, and monitored for adverse events or toxicities, immediately following dosing, and again at 30 days.
  Interventions: Drug: Intravenous Infusion of UCLSCs

INTERVENTIONS:
Drug: Intravenous Infusion of UCLSCs — The first 3 subjects will be administered 50 x 10^6 ULSCs reconstituted in PBS with 1% human serum albumin in a volume of 250 ml, and monitored for adverse events or toxicities, immediately following dosing, and again at 30 days.

SUMMARY:
This is a Phase I, single ascending dose, first in human, open-label, non-controlled, dose-escalation trial that will investigate intravenous infusions of Umbilical cord lining stem cells (UCLSCs) in Left Ventricular Assist Device (LVAD) patients.

This study will recruit patients from the Advanced Heart Failure and LVAD Clinic at the University of Florida, including recently implanted patients, as well as patients on chronic long-term support, with the goal of enrolling up to 9 subjects to participate in the study.

DETAILED DESCRIPTION:
Subjects will be entered into a 3+3 dose escalation study, a standard design for initial trials to evaluate tolerability of a therapeutic agent and identify a maximal tolerated dose if indeed toxicities are identified in the pre-specified dosing range. The first 3 subjects will be administered 50 x 10^6 ULSCs reconstituted in PBS with 1% human serum albumin in a volume of 250 ml, and monitored for adverse events or toxicities, immediately following dosing, and again at 30 days. Safety endpoints will be reviewed by the DSMB and depending on the response, the dose will be escalated to 100 x 10^6 and 200 x 10^6 ULSC in a constant 250 ml volume. We will enroll only 9 subjects in the case that no subject experiences toxicity, only expanding the cohort in the event that a subject experiences toxicity at a particular dose.

This specific dose escalation approach is based on the following considerations:

There is not yet a standard dosing regimen for cell therapy in heart failure patients. The previous MSC trial in LVAD patients provided 150 million cells. The RIMECARD trial (Bartolucci et al, Circ Res 2017 Oct 27;121(10):1192-1204. PMID 28974553) provided umbilical cord-derived MSC for patients with heart failure via intravenous infusions of 1x106 cells/kg. Similarly, another Phase IIa trial of MSCs in HFrEF used 1.5x106 cells/kg (Butler et al., Circ Res 2017 Jan 20;120(2):332-340. PMID 27856497). Since our LVAD patients range in size from 50 to > 100kg, we believe the selected range of doses is reasonable for this patient population.

In addition, in ongoing studies in COVID 19 ARDS, IND# 19979, we have provided 100 x 106 ULSCs with no adverse safety signals. Moreover, in our non-clinical animal models, we demonstrated safety at doses ranging from a high dose of 1 x 106 cells/mouse, which is equivalent to approximately 5 x 107 cells/kg in humans and a low dose of 5 x 104 cells/mouse which is equivalent to approximately 2.5 x 106 cells/kg in humans. The dose tested in the high dose preclinical study would scale to administration of over 2.5 billion cells in an individual weighing 100 pounds.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age
2. Have heart failure with reduced ejection fraction and a durable centrifugal flow LVAD
3. Be on a stable regimen of heart failure medications for at least two weeks, including ACE/ARB/ARNi unless there is a documented contraindication to their use. These medications will be provided at an optimized, guideline-directed maximally tolerated dose.

Exclusion Criteria:

1. Durable Biventricular support
2. An axial flow LVAD
3. History of Crohn's Disease, Ulcerative Colitis, or other Inflammatory Bowel Disease on active treatment
4. LVAD implantation within the last 30 days
5. Anticipated need for non-cardiac surgery within the next 12 months
6. Evidence of active systemic infection at time of study product delivery
7. Evidence of infectious diseases such as hepatitis B, hepatitis C and HIV
8. Prior heart transplant recipients
9. Active cancer (or prior diagnosis of cancer within the past 2 years)
10. Recent (<14 days) or active use of immunosuppressive drugs (including but not limited to high-dose corticosteroids [>1 mg/kg of prednisone equivalent], TNF-α blockers, cyclosporine) not including NSAIDs or corticosteroids used for IV dye allergy only)
11. Chronic auto-immune or auto-inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
12. Recent or planned use of vaccination with live attenuated viruses within the next 30 days
13. Allergy to rubber or latex, or to DMSO.
14. Pregnancy or breastfeeding; fertile women must use contraception to avoid pregnancy.
15. Patient has known hypo- or hyper-coagulable state such as disseminated intravascular coagulation and heparin induced thrombocytopenia (HIT)
16. Platelet count < 100K
17. Inability to maintain an INR of 2-3
18. Inability to give informed consent
19. Cognitive or language barriers that prohibit obtaining informed consent or any study elements (interpreter permitted)
20. Any other condition that, in the judgment of the Investigator, would be a contraindication to enrollment, study product administration, or follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Dose Limiting Toxicity (DLT) that begins during or following ULSC infusion | Within 24 hours
  Dose Limiting Toxicities are treatment-emergent suspected adverse reactions graded severe, such as severe infusion-related hypersensitivity toxicities of grade ≥3, and any serious adverse event (SAE). (Note: DLT during an infusion will stop that infusion in that subject.)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ahmed, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed MM, Meece LE, Handberg EM, Pepine CJ. Intravenous administration of umbilical cord lining stem cells in left ventricular assist device recipient: Rationale and design of the uSTOP LVAD BLEED pilot study. Am Heart J Plus. 2022 May 8;16:100142. doi: 10.1016/j.ahjo.2022.100142. eCollection 2022 Apr. PMID 38559284